CLINICAL TRIAL: NCT06845722
Title: Combined Effects of Balance and Cognitive Training on Executive Functions, Balance and Quality of Life in Patients With Multiple Sclerosis
Brief Title: Combined Effects of Balance and Cognitive Training in Patients With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0249
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: balance; cognitive training; executive function; quality of life; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Balance Training + Cognitive Rehabilitation) (Experimental): Group A will receive both balance training and cognitive rehabilitation twice a week for 12 weeks and each session will last for 1 hour.
  Interventions: Other: Balance training; Other: Cognitive Rehabilitation:
- (Balance Training) (Active Comparator): Group B will receive only balance training twice a week for 12 weeks and each session will last for 1 hour.
  Interventions: Other: Balance training

INTERVENTIONS:
Other: Balance training — * The balance training will be given for 12 weeks (2 sessions/week, 30-35 in each) that included six balance exercises per training session.
  * After 5-min warm-up program including general (e.g., neck rolls, shoulder circles, side bends, hip circles, marsh in place) and specific (e.g., two-/one-legged stance on unstable devices, forward/backward beam walking).
  * Two sets per balance exercise will be performed for 30s each with a 60s rest period between sets and a 90 s break between exercises. Yet, both groups will execute the same training volume (i.e., number of exercises, number of sets per exercise, and duration per set of exercise).
  * Progression during training will be achieved by means of increasing exercise duration (i.e., from 30s over 45s to 60 s), change of stance (i.e., two-legged stance, tandem. stance, one-legged stance) and walking (i.e., forward, backward) condition, manipulation of visual input (e.g., eyes opened vs. closed), and concurrent execution of cognitive
Other: Cognitive Rehabilitation: — * The cognitive rehabilitation will be given for 12 weeks ( 2 sessions/week,30 min each session). The individual sessions for the CR approach will involve an individualized intervention focusing on a personally meaningful goal (e.g., maintaining attention while flipping cards and finding matching pairs, learning to use a cellular phone, remembering the names of people).
  * The individual sessions will be consisted of practical strategies and aids, compensation strategies (e.g., using a memory notebook), and the techniques for stress management to improve performance and functioning in relation to goals. The group sessions of CR involved some tasks of cognitive training.
  * The group sessions will be focused on practicing time-and-place orientation through paper-and pencil tasks provided by a therapist and use of a calendar and personal memory notebook or cellular phone at the start of each session. (30)
  * The group sessions also involved matching faces and names and learning memory
  Arms: (Balance Training + Cognitive Rehabilitation)

SUMMARY:
Multiple sclerosis is a potentially disabling disease of the brain and spinal cord involving the central nervous system. Multiple Sclerosis can cause balance and cognitive impairment in patients, affecting overall quality of life. Balance and cognitive training can effectively improve the overall executive function and mobility in patients with multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis is a potentially disabling disease of the brain and spinal cord involving the central nervous system. Multiple Sclerosis can cause balance and cognitive impairment in patients, affecting overall quality of life. Balance and cognitive training can effectively improve the overall executive function and mobility in patients with multiple sclerosis. Enhancing cognitive abilities and balance skills in MS patients can be accomplished through cognitive rehabilitation that prioritizes processing speed. In MS patients, this kind of intervention can also delay the onset of secondary cognitive deficits. This study aims to investigate the combined effects of balance and cognitive training on executive functions, balance, and quality of life in patients with multiple sclerosis.

The randomized controlled trial will be carried out at multi-settings in Lahore in 10 months after the approval of synopsis. The total 42 participants meeting the inclusion criteria will be included in this study through a non-probability convenience sampling technique. Participants will be randomly assigned into 2 groups using computer generated method. Group A and Group B participants both will receive balance training, while Group A participants will also receive cognitive training twice a week for 12 weeks and each session will last for 1 hour. Outcome measure tools will be Montreal cognitive assessment (MOCA) for cognitive assessment, Berg balance scale BBS for balance assessment and SF36 questionnaire for assessment of quality of life. The data will be collected at baseline and post treatment to measure the outcome measures. Data will be analyzed by SPSS version 26. Statistical significance will be set at p=0.05. The normality of data will be checked by using Shapiro-Wilk test. For the between group analysis of parametric data, Independent T test will be used, while for within group analysis Paired T test will be used. Kruskal-Wallis test will be applied for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patients should be 40-55 years.(20)
* Gender: both males and females
* Patients with diagnosed multiple sclerosis.
* According to MOCA assessment, patients with scoring 21-25 will be included. (Patients with executive function deficits due to Multiple Sclerosis including relapsing-remitting, primary progressive and secondary progressive MS).(21)
* Patients feel difficulty in Impaired Balance and walking.
* According to the Berg Balance Scale, patients under 21-45 will be included.(22)

Exclusion Criteria:

* Participants with a history of moderate to severe head injury, stroke and seizures will be excluded(23)
* Cognitive impairment due to presence of current or past neurological disorders other than Multiple Sclerosis will be excluded.(23)
* Participants with active major psychiatric illness (such as schizophrenia, bipolar disorder or depressive disorder) will be excluded(23)
* Patients with history of learning disabilities, severe head trauma, alcohol or drug abuse will be excluded(23)

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
I. Montreal Cognitive Assessment for Cognitive Impairment: | 12 Weeks
  • For Cognitive Impairment: This outcome measurement tool will be used for assessment of cognitive impairment. In patients with multiple sclerosis.MoCA is a screening instrument that evaluates seven cognitive domains on a single page and scores range from 0 to 30. The domains are: visuospatial/executive functions, naming, verbal memory registration and learning, attention, abstraction, 5-minute delayed verbal memory, and orientation.(24) The MoCA scoring suggested a cutoff score of 26, with those scoring 25 or below suspected of having (MCI).(24)MoCA had demonstrated an excellent diagnostic validity of 0.89 (95% CI: 0.83-0.95)(25).The inter-rater reliability or an ICC value of MoCA was 0.96 (95% CI: 0.91-0.98.
II. Berg Balance Scale for balance assessment: | 12 Weeks
  • For Balance assessment: This outcome measurement tool will be used for assessment of Balance in patients with multiple sclerosis. The BBS contains 14 static and dynamic balance activities related to daily life. The BBS tasks progress in challenges: from sitting to standing, standing with narrow base of support, and finally to tandem and single-leg stance. Scoring is on a 5-point ordinal scale with 0 indicating an inability to complete the task and 4 as independent with completing the task.(22).The maximum score of 56 indicates good balance. The scale takes approximately 10 to 20 minutes to complete requiring minimal equipment (chair, stopwatch, ruler, and step) and minimal space.(22)The score of 56 indicates the normal functional balance.(22).The score less than 45 will indicates the higher risk of fall due to impaired balance.(22).The validity of the BBS is (7 = -0.50, P <.001,4 and r = -0.58, P < 005).(26).BBS had strong test-retest reliability (ICC = 0.90).26

SECONDARY OUTCOMES:
III. Short form of SF 36-Item health survey for Quality of life: | 12 Weeks
  • For assessment of Quality of life: A 36-item short-form (SF-36) was constructed to survey health status and quality of life. The SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. The survey is constructed for self-administration by persons 14 years of age and older, and for administration by a trained therapist as well.(27).The items are categorized, totaled, and converted into a scale ranging from 0 (the worst condition of health) to 100

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad M.Phill, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schedler S, Tenelsen F, Wich L, Muehlbauer T. Effects of balance training on balance performance in youth: role of training difficulty. BMC Sports Sci Med Rehabil. 2020 Nov 23;12(1):71. doi: 10.1186/s13102-020-00218-4. PMID 33292455
- [Background] Carson N, Leach L, Murphy KJ. A re-examination of Montreal Cognitive Assessment (MoCA) cutoff scores. Int J Geriatr Psychiatry. 2018 Feb;33(2):379-388. doi: 10.1002/gps.4756. Epub 2017 Jul 21. PMID 28731508
- [Background] Gil-Gonzalez I, Martin-Rodriguez A, Conrad R, Perez-San-Gregorio MA. Quality of life in adults with multiple sclerosis: a systematic review. BMJ Open. 2020 Nov 30;10(11):e041249. doi: 10.1136/bmjopen-2020-041249. PMID 33257490
- [Background] Azimian M, Yaghoubi Z, Ahmadi Kahjoogh M, Akbarfahimi N, Haghgoo HA, Vahedi M. The Effect of Cognitive Rehabilitation on Balance Skills of Individuals with Multiple Sclerosis. Occup Ther Health Care. 2021 Jan;35(1):93-104. doi: 10.1080/07380577.2021.1871698. Epub 2021 Jan 12. PMID 33433260
- [Background] Arntzen EC, Braaten T, Fikke HK, Normann B. Feasibility of a new intervention addressing group-based balance and high-intensity training, physical activity, and employment in individuals with multiple sclerosis: a pilot randomized controlled trial. Front Rehabil Sci. 2024 Jan 8;4:1258737. doi: 10.3389/fresc.2023.1258737. eCollection 2023. PMID 38259873
- [Background] Perucca L, Scarano S, Russo G, Robecchi Majnardi A, Caronni A. Fatigue may improve equally after balance and endurance training in multiple sclerosis: a randomised, crossover clinical trial. Front Neurol. 2024 Jan 19;15:1274809. doi: 10.3389/fneur.2024.1274809. eCollection 2024. PMID 38385033
- [Background] Feinstein A, Amato MP, Brichetto G, Chataway J, Chiaravalloti ND, Cutter G, Dalgas U, DeLuca J, Farrell R, Feys P, Filippi M, Freeman J, Inglese M, Meza C, Motl RW, Rocca MA, Sandroff BM, Salter A; CogEx Research Team. Cognitive rehabilitation and aerobic exercise for cognitive impairment in people with progressive multiple sclerosis (CogEx): a randomised, blinded, sham-controlled trial. Lancet Neurol. 2023 Oct;22(10):912-924. doi: 10.1016/S1474-4422(23)00280-6. PMID 37739574
- [Background] Henry A, Lannoy S, Chaunu MP, Tourbah A, Montreuil M. Social cognition and executive functioning in multiple sclerosis: A cluster-analytic approach. J Neuropsychol. 2022 Mar;16(1):97-115. doi: 10.1111/jnp.12248. Epub 2021 May 14. PMID 33989458
- [Background] Lassmann H, Bruck W, Lucchinetti CF. The immunopathology of multiple sclerosis: an overview. Brain Pathol. 2007 Apr;17(2):210-8. doi: 10.1111/j.1750-3639.2007.00064.x. PMID 17388952
- [Background] Graves JS, Krysko KM, Hua LH, Absinta M, Franklin RJM, Segal BM. Ageing and multiple sclerosis. Lancet Neurol. 2023 Jan;22(1):66-77. doi: 10.1016/S1474-4422(22)00184-3. Epub 2022 Oct 7. PMID 36216015
- [Background] Marcus R. What Is Multiple Sclerosis? JAMA. 2022 Nov 22;328(20):2078. doi: 10.1001/jama.2022.14236. PMID 36413229